CLINICAL TRIAL: NCT06690450
Title: A Randomized Study to Assess the Safety and Tolerability of 200mg and 100mg of Venofer Administered to Hemodialysis (HD) Patients
Brief Title: Safety and Tolerability of 200mg and 100mg of Venofer Administered to Hemodialysis(HD) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1VEN01015
Record Dates: First submitted 2019-02-07; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Hemodialysis
MeSH Terms: interventions — Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Venofer® 200 mg (Experimental): A single 200 mg dose of Venofer® administered by slow intravenous push over 5 minutes.
  Interventions: Drug: Venofer® 200 mg
- Venofer® 100 mg (Active Comparator): A single 100 mg dose of Venofer® administered by slow intravenous push over 2 minutes without a test dose
  Interventions: Drug: Venofer® 100 mg

INTERVENTIONS:
Drug: Venofer® 200 mg — A single 200 mg dose of Venofer® administered by slow intravenous push over 5 minutes
  Other Names: Iron sucrose
  Arms: Venofer® 200 mg
Drug: Venofer® 100 mg — A single 100 mg dose of Venofer® administered by slow intravenous push over 2 minutes without a test dose.
  Other Names: Iron sucrose
  Arms: Venofer® 100 mg

SUMMARY:
The Objective of this study is to assess the Safety and Tolerability of 200 mg and 100 mg of Venofer Administered to Hemodialysis(HD) Patients.

DETAILED DESCRIPTION:
This is a randomized open label multi-center study of two parallel patient groups undergoing hemodialysis. Group A will receive 200 mg of iron sucrose, while Group B will receive 100 mg of iron sucrose during the study. The duration of the study for each patient will be approximately 3 weeks including a screening phase, a treatment visit and a follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Males or females over 18 years of age and able to give informed consent.
* Undergoing hemodialysis.
* If receiving epoetin α, then the dose was stable.
* Percentage serum transferrin saturation (TSAT) <50% and serum ferritin <800 ng/mL.
* Absence of infection, malignancy, or surgery in the month prior to study start.
* Intolerance of other iron products did not preclude participation in this study.

Exclusion Criteria:

* Known sensitivity to any component of Venofer®.
* Suffering from concomitant severe diseases of the liver, cardiovascular system, severe psychiatric disorders or other conditions which, in the opinion of the investigator, made participation unacceptable.
* Serious bacterial, viral infection, or other acute infectious illness (e.g., hepatitis) unless completely resolved at least 4 weeks prior to inclusion in the study.
* Pregnancy or lactation.
* HIV positive by medical history or laboratory test (optional), or active hepatitis.
* Anemia caused by diseases (including systemic lupus erythematosus (SLE), rheumatoid arthritis, myeloma, or hereditary hemoglobinopathies) other than chronic renal failure or iron deficiency.
* Asthma.
* Clinical evidence of gastrointestinal bleeding.
* Would probably require blood transfusion or might undergo a renal transplant during the study.
* Anticipated surgery of any kind during the study other than vascular access surgery.
* Received an investigational drug within 30 days prior to screening.
* Previously participated in another Venofer® study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2001-08 (Actual); Primary Completion 2002-01 (Actual); Study Completion 2002-02 (Actual)

PRIMARY OUTCOMES:
The number of participants with treatment-emergent adverse events (TEAEs) as assessed by CTCAE v4.0 | 3 to 6 days
  Any untoward medical events were elicited by nonspecific questions such as "Have you noticed any problems".

SECONDARY OUTCOMES:
The number of participants prematurely discontinued the study due to an adverse event | 3 to 6 days
  The investigator determined whether any adverse event warranted removal of a subject from the study

CONTACTS AND LOCATIONS:
Overall Officials: Carol Duffy, D.O.,FACC, Study Director — Medical Director